CLINICAL TRIAL: NCT04083118
Title: Non-invasive Detection of Bicuspid Aortic Valve-Related Thoracic Aortopathy
Brief Title: Assessment of Risk in Thoracic Aortopathy Using 18F-Sodium Fluoride
Acronym: AoRTAS
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/0261; FS/19/15/34155 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2019-09-02; First posted 2019-09-10 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Bicuspid Aortic Valve; Thoracic Aortic Aneurysm; Aortic Dissection
Keywords: positron emission tomography; sodium fluoride; bicuspid aortic valve; thoracic aortic aneurysm; aortopathy
MeSH Terms: conditions — Bicuspid Aortic Valve Disease; Aortic Aneurysm, Thoracic; Aortic Dissection | interventions — Physical Examination; Pulse Wave Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples taken at each visit with ethical approval and consent to store for DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bicuspid aortic valve: 80 patients with bicuspid aortic valve with or without an aortic aneurysm
  Interventions: Diagnostic Test: clinical evaluation, blood markers, pulse wave analysis, 18F sodium fluoride PET/CT and PET/MRI; Diagnostic Test: Repeat 18F sodium fluoride PET/MRI
- controls: 20 healthy volunteer controls age and sex matched to 20 of the bicuspid aortic valve patients
  Interventions: Diagnostic Test: clinical evaluation, blood markers, pulse wave analysis, 18F sodium fluoride PET/CT and PET/MRI

INTERVENTIONS:
Diagnostic Test: clinical evaluation, blood markers, pulse wave analysis, 18F sodium fluoride PET/CT and PET/MRI — Patients will receive a structured clinic history, examination, blood sampling, pulse wave analysis, pulse wave velocity, 18F-sodium fluoride PET/CT, 18F-sodium fluoride PET/MRI with detailed cardiac magnetic resonance imaging and magnetic resonance imaging of the aorta
Diagnostic Test: Repeat 18F sodium fluoride PET/MRI — as per first study visit but without the PET/CT
  Groups: Bicuspid aortic valve

SUMMARY:
Patients with bicuspid aortic valve-related aortopathy are at increased risk of aortic dilatation, dissection and rupture. Currently, risk stratification is largely based on aortic diameter measurements, with those deemed high risk referred for aortic replacement surgery. This approach is imperfect, and potentially exposes many patients to unnecessary high-risk aortic surgery, or fails to identify those at risk of dissection or rupture with smaller diameters. In patients with abdominal aortic aneurysms, the investigators recently demonstrated that uptake of 18F-sodium fluoride predicts disease progression and clinical events independent of aneurysm diameter and standard clinical risk factors. Based on the investigators preliminary data, a study was proposed to look at 18F-sodium fluoride uptake in patients with bicuspid aortic valve-related aortopathy. The proposed study will shed light on the underlying pathological processes involved in aortic complications of this disease as well as potentially providing an important risk marker to predict disease progression and guide the need for major aortic surgery.

DETAILED DESCRIPTION:
Bicuspid aortic valve, along with other congenital conditions affecting the aortic wall, has been associated with elastic fibre loss, decrease in size of elastic lamellae, increased collagen deposition and smooth muscle loss compared to healthy controls on both light microscopy and electron microscopy. Further, analysis of site specific regions of the ascending aorta using biopsy specimens demonstrated significant differences in the apoptosis rate and survival of smooth muscle cells favouring the lesser curvature over the greater curvature of the aorta (the area of greater wall shear stress).

Studies to date suggest vessel wall microcalcification (lesions<50μm) is a dynamic marker of this vessel wall pathology: the end-product of a pathological process involving vessel wall inflammation, apoptosis and necrosis of medial smooth muscle cells and subsequent elastic fibre degradation. Granular medial calcinosis, the deposition of microcalcification in the medial layer of resected aortic tissue, has been recognised as a significant feature of bicuspid aortic valve-related aortopathy when compared to aortic samples taken from patients with tricuspid valves.

Recent histological analysis of human and murine Marfan aortas demonstrated elastin breaks co- localising with areas of microcalcification in aortic media. Further, the areas of elastin break were significantly correlated to decreased distensibility and increased aortic diameter. Finally, the group demonstrated an elastin receptor complex-ERK1/2-ALP-mediated mechanism for increased microcalcification deposition. Although focused on Marfan syndrome, these results are relevant to bicuspid aortic valve-related aortopathy as they suggest microcalcification is associated with elastic fibre breakdown, a proposed mechanism of bicuspid aortic valve aneurysm formation at areas of high wall shear stress. The ability to demonstrate and quantify aortic microcalcification, both ex vivo and non-invasively in vivo in patients with bicuspid aortic valve-related aortopathy would be important step in improving our knowledge of the pathological process underpinning this condition.

Positron emission tomography (PET) utilises a radiotracer which provides functional information on tissues at the cellular or molecular level. Because of its limited spatial resolution, PET images are combined with computed tomography (CT) or magnetic resonance imaging (MRI) so that the functional PET images can be co-registered with the detailed anatomical and structural images afforded by CT or MRI. While CT or MRI alone has been utilised in a wide range of cardiovascular diseases and can identify larger areas of macrocalcification (>200 μm), PET/CT using 18F-sodium fluoride has been used to identify vessel wall microcalcification (calcific lesions <50 μm) that is not detectable on CT or MRI. 18F-Sodium fluoride has been extensively validated as a radiotracer of microcalcification utilising electron microscopy, immunohistochemical analysis, pharmacodynamic concentration-response curves, and ex vivo and in vivo micro-PET/CT on vessel wall sections. 18F-Sodium fluoride uptake is mediated through exchange of fluoride ions with hydroxyl groups of hydroxyapatite, the major constituent of vessel wall calcification. Positron emission tomography using 18F-sodium fluoride has demonstrated significant promise as identifying active vessel wall pathology in a number of cardiovascular diseases including carotid, coronary, aortic valve, and abdominal aortic aneurysm disease. The use of 18F-sodium fluoride PET imaging in thoracic aortic aneurysms is novel.

There is a correlation between areas of high wall stress and intimal tear location location. Further, aneurysmal aortic tissue has been demonstrated to have reduced delamination strength in both longitudinal and circumferential dimensions: evidence for an involvement of haemodynamic effects on precipitating dissection. Time resolved 3D blood flow captured on MRI, also known as 4D-flow MRI, is an evolving research tool which non-invasively captures patient-specific regionalised blood flow and velocity, allowing calculation of aortic wall sheer stress, and has been used to study bicuspid aortic valve-related aortopathy. A study pairing pre-operative 4D-flow MRI and post-operative biopsies of aortic tissue have demonstrated a decrease in elastin at sites of high aortic wall stress, suggesting a relationship between haemodynamics and the structural composition of the aneurysmal aortic wall. The ability to demonstrate a pathological process associated with aneurysmal weakness could be an important step to better identifying high risk lesions.

ELIGIBILITY:
Inclusion Criteria:

* Bicuspid aortic Valve or Age-sex matched healthy volunteer

Exclusion Criteria:

* Pregnancy
* eGFR < 30
* previous aortic replacement surgery
* previous aortic valve surgery
* contrast allergy
* other reason unable to undergo MRI

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with bicuspid aortic valve and a variety of ascending aortic sizes
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-09-03 (Actual); Study Completion 2023-09-03 (Actual)

PRIMARY OUTCOMES:
Aortic growth rate | At 1-2 years after baseline visit
  Correlate baseline 18F sodium fluoride PET uptake with aortic growth rate, a marker of aortic wall remodelling, over 1-2 years

SECONDARY OUTCOMES:
Aortic stiffness | 1-2 years (at second study visit)
  Aortic stiffness, which is a biomechanical marker of how elastic the aortic wall is, has been associated with increased aortic event rates in patients with connective tissue disorders. We will measure aortic stiffness using a variety of metrics including distensibility, elastic modulus, stiffness index (all MRI derived) and pulse wave velocity (deprived using application tomography). The change in aortic stiffness and baseline aortic stiffness will be correlated with baseline PET
Wall shear stress | 1 year (at baseline visit)
  Wall shear stress is extrapolated from 4D MRI and is proposed to be linked with histological changes in the aortic wall as well as increased dilatation. We will compare areas of high wall shear stress to those of high PET uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J Fletcher, MD, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fletcher AJ, Nash J, Syed MBJ, Macaskill MG, Tavares AAS, Walker N, Salcudean H, Leipsic JA, Lim KHH, Madine J, Wallace W, Field M, Newby DE, Bouchareb R, Seidman MA, Akhtar R, Sellers SL. Microcalcification and Thoracic Aortopathy: A Window Into Disease Severity. Arterioscler Thromb Vasc Biol. 2022 Aug;42(8):1048-1059. doi: 10.1161/ATVBAHA.122.317111. Epub 2022 Jun 30. PMID 35770666
- [Background] Fletcher AJ, Lembo M, Kwiecinski J, Syed MBJ, Nash J, Tzolos E, Bing R, Cadet S, MacNaught G, van Beek EJR, Moss AJ, Doris MK, Walker NL, Dey D, Adamson PD, Newby DE, Slomka PJ, Dweck MR. Quantifying microcalcification activity in the thoracic aorta. J Nucl Cardiol. 2022 Jun;29(3):1372-1385. doi: 10.1007/s12350-020-02458-w. Epub 2021 Jan 20. PMID 33474695
- See also: BHF website — https://europepmc.org/grantfinder/grantdetails?query=pi%3A%22Walker%2BN%22%2Bgid%3A%22FS%2F19%2F15%2F34155%22%2Bga%3A%22British+Heart+Foundation%22
- See also: University of Edinburgh website — https://www.ed.ac.uk/clinical-sciences/edinburgh-imaging/news/2019-news/07-mar-19-aortas-study